CLINICAL TRIAL: NCT05953792
Title: Selecting the Vertebra Above Sagittal Stable Vertebra as the Distal Fusion Level in Scheuermann's Kyphosis
Brief Title: Selecting the SSV-1 as LIV in Scheuermann's Kyphosis
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-LCYJ-DBZ-05
Record Dates: First submitted 2023-07-02; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Scheuermann's Kyphosis
MeSH Terms: conditions — Scheuermann Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thoracic kyphosis: patients with their kyphotic apex located at T10 or above
  Interventions: Procedure: Select the vertebra above sagittal stable vertebra as the distal fusion level
- thoracolumbar kyphosis: patients with their kyphotic apex located below T10
  Interventions: Procedure: Select the vertebra above sagittal stable vertebra as the distal fusion level

INTERVENTIONS:
Procedure: Select the vertebra above sagittal stable vertebra as the distal fusion level — The surgeries were performed by the same surgical team. Multi-level Ponte osteotomies were performed across the apex of the kyphosis after complete exposure of the spine, with resection of supra- and inter-spinous ligaments, ligamentum flavum, and the whole facet joints. After placement of the pedicle screws at the expected fusion levels, pre-contoured rods were attached to the screws followed by segmental compression. During rod placement, two to three rounds of compression in the area with Ponte osteotomies were employed to enhance kyphosis correction. Satellite rods were routinely added to long rods and implanted with duet screws. The final tightening was performed, and the posterior fusion was completed with a mixture of local and allogeneic bone. Due attention was given to preserving the posterior ligamentous structures at the upper and lower junctional areas.

SUMMARY:
The proper selection of the lowest instrumented vertebra (LIV) remains controversial in the surgical treatment of Scheuermann's disease and there is a paucity of studies investigating the clinical outcomes of fusion surgery when selecting the vertebra one level proximal to the sagittal stable vertebra (SSV-1) as LIV. The purpose of this study is to investigate whether SSV-1 could be a valid LIV for Scheuermann kyphosis (SK) patients with different curve patterns.

DETAILED DESCRIPTION:
The proper selection of the lowest instrumented vertebra (LIV) remains controversial in the surgical treatment of Scheuermann's disease and there is a paucity of studies investigating the clinical outcomes of fusion surgery when selecting the vertebra one level proximal to the sagittal stable vertebra (SSV-1) as LIV. The purpose of this study is to investigate whether SSV-1 could be a valid LIV for Scheuermann kyphosis (SK) patients with different curve patterns.

This was a prospective study on consecutive SK patients treated with posterior surgery between January 2018 and September 2020, in which the distal fusion level ended at SSV-1. The LIV was selected at SSV-1 only in patients with Risser > 2 and with LIV translation less than 40mm. All of the patients had a minimum of 2-year follow-up. Patients were further grouped based on the sagittal curve pattern as thoracic kyphosis (TK) and thoracolumbar kyphosis (TLK). Radiographic parameters including global kyphosis (GK), lumbar lordosis (LL), sagittal vertical axis (SVA), LIV translation, pelvic incidence (PI), pelvic tilt (PT), sacral slope (SS) were measured preoperatively, postoperatively and at the latest follow-up. The intraoperative and postoperative complications were recorded. The Scoliosis Research Society (SRS)-22 scores were performed to evaluate clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SK patients;
* underwent one-stage posterior spinal fusion (PSF) with multi-level Ponte osteotomies;
* selecting SSV-1 as LIV;
* with a minimum follow-up of 2 years.

Exclusion Criteria:

* with previous spinal surgical history;
* with any other spinal deformities;
* without complete follow-up data.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 36 SK patients (including 23 with TK and 13 patients with TLK) were included in this study, among which 29 were male, and 7 were female.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Global kyphosis (GK) in degrees | 24 months
  Measured on anteroposterior and lateral radiographs and defined as the angle from upper to lower most tilted end vertebrae.
Lumbar lordosis (LL) in degrees | 24 months
  Measured on anteroposterior and lateral radiographs and defined as the angle between the the superior end plate of L1 and S1
Sagittal vertical axis (SVA) in millimeters | 24 months
  Measured on anteroposterior and lateral radiographs and defined as the horizontal distance between C7PL and the posterior superior corner of sacrum.

SECONDARY OUTCOMES:
Rates of distal junctional kyphosis | 24 months
  record the incidence of the distal junctional kyphosis at the last follow-up. Distal junctional kyphosis was defined as a distal junctional angle ≥10˚, or a distal junctional angle ≥ 10˚ than the preoperative measurement
Scoliosis Research Society (SRS)-22 questionnaire | 24 months
  The Scoliosis Research Society (SRS)-22 questionnaire is adopted to assess the patient-reported outcomes. The overall score can range from 22 to 110 points, and higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No